CLINICAL TRIAL: NCT05889247
Title: Circulating Tumor DNA Guided Treatment Monitoring in Advanced Lung Cancer - a Randomized Interventional Study
Brief Title: Circulating Tumor DNA Guided Treatment Monitoring in Advanced Lung Cancer
Acronym: PRELUCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Malene Støchel Frank, Medical Oncologist, PhD, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-1011
Record Dates: First submitted 2023-05-08; First posted 2023-06-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: liquid biopsy; treatment monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA monitoring (Experimental): Treatment monitoring by longitudinal circulating tumor DNA measurements and Quality of Life assessments
  Interventions: Other: Circulating tumor DNA treatment monitoring
- CT scan monitoring (No Intervention): Treatment monitoring by longitudinal CT scans (standard) and Quality of Life Assessments

INTERVENTIONS:
Other: Circulating tumor DNA treatment monitoring — A comparison of treatment monitoring by circulating tumor DNA and CT scans (standard) in patients with newly diagnosed advanced Non-Small Cell Lung Cancer (NSCLC)
  Other Names: Quality of Life assessments
  Arms: ctDNA monitoring

SUMMARY:
The study is a prospective randomized interventional study including patients with advanced non-small cell lung cancer, receiving immunotherapy, with the aim of optimizing treatment monitoring. The study aims to investigate the clinical utility of liquid biopsy monitoring in order to reduce the numbers of inefficient treatments and needless toxicity - and to explore the cost-effectiveness and cost-utility of introducing liquid biopsy monitoring in daily clinical practice.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death worldwide with Non-Small Cell Lung Cancer (NSCLC) being the most common subtype. Performance status deterioration due to progressive symptoms and toxicity by treatments are major challenges in managing advanced NSCLC patients. Moreover, standard treatment monitoring by radiologic scans is often imprecise. This technology has limited sensitivity as only a visible increase or decrease in tumor mass can be evaluated, making interpretation challenging and conclusions of whether patients benefit from treatment indefinite. Interpretation of radiologic scans has been further challenged after implementation of immunotherapy, causing immunotherapy-induced recruitment of immune cells resembling increment in tumor size, called "pseudo-progression." More sensitive methods are highly needed to reduce ineffective treatments and needless toxicity. Liquid biopsy has the potential to overcome these challenges by measuring molecular changes with high precision in a dynamic manner. Recent studies have demonstrated its promising potential as a biomarker predictive of treatment efficacy and overall survival. In a recent real-life study, investigators found that ctDNA measurements could reduce 33% of likely inefficient treatments and clarify 79% of non-conclusive CT-scans, highlighting the clinical potential. A randomized interventional multicenter study will be performed, investigating the true clinical potenial of liquid biopsy compared to standard monitoring by radiological scans. A total of 350 patients with advanced NSCLC will be included in the study from three Departments of Clinical Oncology. In the interventional arm, liquid biopsy monitoring will be the basis for treatment discontinuation before the standard two years of immunotherapy in patients reaching a complete molecular response in plasma. Thus clarifying the question if treatment duration can be reduced for the benefit of patients and health cost.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically verified, Non-Small Cell Lung Cancer (NSCLC)
* Advanced or locally advanced disease without curative intended treatment options
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) score of Performance Status (PS) 0-1
* Measurable disease according to the iRECIST criteria version 1.1.
* Eligible to first line immunotherapy (monotherapy)
* Signed informed consent

Exclusion Criteria:

* Targetable alterations in EGFR, ALK or ROS-1
* Other active cancers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 3 years
  Overall Survival

SECONDARY OUTCOMES:
Physicians Global Assessment to measure quality of life | through study completion, an average of 3 years
  Physicians Global Assessment to measure quality of life
Common Terminology Criteria for Adverse Events | through study completion, an average of 3 years
  Common Terminology Criteria for Adverse Events
Number of Treatments | From randomization to first detection of progressive disease, an average of 3 years
  Number of treatments given and not given
Health Cost/Utility | From randomization to first detection of progressive disease, an average of 3 years
  A health cost and utility analysis of patients in both arms

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Department of Clinical Oncology, Hillerød, Region H
  - Department of Clinical Oncology and Palliative Care, Næstved, Region Sjælland
  - Department of Clinical Oncology and Palliative Care, Roskilde, Region Sjælland
  - Department of Oncology, Aalborg
  - Department of Oncology, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen ME, Nyhus CH, Szejniuk WM, Wahlstrom S, Timm S, Pallisgaard N, Madsen MG, Mikkelsen MD, Ahlborn LB, Gehl J, Frank MS. ctDNA guided immunotherapy in patients with advanced non-small cell lung cancer: a nationwide Danish, randomised, intervention study (PRELUCA-PRediction in LUng CAncer Treatment) - study protocol. BMJ Open. 2026 Feb 2;16(2):e100311. doi: 10.1136/bmjopen-2025-100311. PMID 41628935